CLINICAL TRIAL: NCT06582732
Title: Prospective, Non-Randomized, Open-Label, Single Center Study to Evaluate the Performance of the Travoprost Intraocular Implant
Brief Title: Performance of the Travoprost Intraocular Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDOS-402-IVIV
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (12-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 12
  Interventions: Drug: Travoprost Intracameral Implant exchanged at Month 12
- Cohort 2 (3-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 3
  Interventions: Drug: Travoprost Intracameral Implant exchanged at Month 3
- Cohort 3 (6-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 6
  Interventions: Drug: Travoprost Intracameral Implant exchanged at Month 6
- Cohort 4 (24-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 24
  Interventions: Drug: Travoprost Intracameral Implant exchanged at Month 24
- Cohort 5 (21-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 21
  Interventions: Drug: Travoprost intracameral implant exchanged at Month 21
- Cohort 6 (18-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 18
  Interventions: Drug: Travoprost intracameral implant exchanged at Month 18
- Cohort 7 (15-month exchange) (Experimental): Travoprost Intracameral Implant Exchanged at Month 15
  Interventions: Drug: Travoprost intracameral implant exchanged at Month 15

INTERVENTIONS:
Drug: Travoprost Intracameral Implant exchanged at Month 12 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 12
  Other Names: iDose TR
  Arms: Cohort 1 (12-month exchange)
Drug: Travoprost Intracameral Implant exchanged at Month 3 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 3
  Other Names: iDose TR
  Arms: Cohort 2 (3-month exchange)
Drug: Travoprost Intracameral Implant exchanged at Month 6 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 6
  Other Names: iDose TR
  Arms: Cohort 3 (6-month exchange)
Drug: Travoprost Intracameral Implant exchanged at Month 24 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 24
  Other Names: iDose TR
  Arms: Cohort 4 (24-month exchange)
Drug: Travoprost intracameral implant exchanged at Month 21 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 21
  Other Names: iDose TR
  Arms: Cohort 5 (21-month exchange)
Drug: Travoprost intracameral implant exchanged at Month 18 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 18
  Other Names: iDose TR
  Arms: Cohort 6 (18-month exchange)
Drug: Travoprost intracameral implant exchanged at Month 15 — intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 15
  Other Names: iDose TR
  Arms: Cohort 7 (15-month exchange)

SUMMARY:
To evaluate the performance of the Travoprost Intracameral Implant by determining residual drug in explanted implants of the Travoprost Intracameral Implant and by determining aqueous humor concentrations of travoprost free acid at specified timepoints post administration through 24 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either open angle glaucoma (i.e. primary, pseudoexfoliation, or pigmentary glaucoma) or ocular hypertenson
* Zero to three topical intraocular pressure lowering medications at the time of Visit 1 (Screening) exam.
* Best spectacle corrected visual acuity of 16 letters or more correctly read at 4 meters or better in each eye.
* Open angle as defined by Shaffer grade ≥ 3 at slit-lamp at the planned implantation site

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle-closure glaucoma; or glaucoma associated with vascular disorders
* Active ocular inflammation, infection or edema
* Clinically significant dystrophy (e.g., bullous keratopathy, Fuch's dystrophy) or clinically significant guttata

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szekely G, Voskanyan LA, Stephens KG, Doan LV, Seal JR, ElMallah MK, Fjield T, Applegate D, Usner DW, Katz LJ, Kothe AC, Navratil T. Aqueous Humor Concentrations of Travoprost Free Acid and Residual Drug in Explanted Implants from Patients Administered a Travoprost Intracameral Implant. Ophthalmol Ther. 2025 May;14(5):989-1003. doi: 10.1007/s40123-025-01130-1. Epub 2025 Mar 24. PMID 40126812

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Initial Study Period
Arm/Group | Cohort 1 (12-month Exchange) | Cohort 2 (3-month Exchange) | Cohort 3 (6-month Exchange) | Cohort 4 (24-month Exchange) | Cohort 5 (21-month Exchange) | Cohort 6 (18-month Exchange) | Cohort 7 (15-month Exchange)
Started | 30; 30 eyes | 30; 30 eyes | 30; 30 eyes | 30; 30 eyes | 30; 30 eyes | 30; 30 eyes | 30; 30 eyes
Completed | 29; 29 eyes | 29; 29 eyes | 28; 28 eyes | 27; 27 eyes | 25; 25 eyes | 29; 29 eyes | 28; 28 eyes
Not Completed | 1; 1 eyes | 1; 1 eyes | 2; 2 eyes | 3; 3 eyes | 5; 5 eyes | 1; 1 eyes | 2; 2 eyes
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 3 | 1 | 2
Not completed — Moved Away | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Post-exchange Study Period
Arm/Group | Cohort 1 (12-month Exchange) | Cohort 2 (3-month Exchange) | Cohort 3 (6-month Exchange) | Cohort 4 (24-month Exchange) | Cohort 5 (21-month Exchange) | Cohort 6 (18-month Exchange) | Cohort 7 (15-month Exchange)
Started | 29; 29 eyes | 29; 29 eyes | 28; 28 eyes | 27; 27 eyes | 25; 25 eyes | 29; 29 eyes | 28; 28 eyes
Completed | 29; 29 eyes | 29; 29 eyes | 28; 28 eyes | 27; 27 eyes | 25; 25 eyes | 29; 29 eyes | 28; 28 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: only a single eye (defined as the study eye) was analyzed in the study
Units Other Than Participants: study eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (12-month Exchange) | Cohort 2 (3-month Exchange) | Cohort 3 (6-month Exchange) | Cohort 4 (24-month Exchange) | Cohort 5 (21-month Exchange) | Cohort 6 (18-month Exchange) | Cohort 7 (15-month Exchange) | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 210
Number analyzed (study eyes) | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 14 | 16 | 14 | 16 | 12 | 103
  >=65 years | 13 | 16 | 16 | 14 | 16 | 14 | 18 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 14 | 15 | 10 | 17 | 16 | 103
  Male | 15 | 14 | 16 | 15 | 20 | 13 | 14 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 210
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Armenia | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 210
Type of Disease [Count of Participants; unit: Participants] — clinical diagnosis of disease type (open angle glaucoma or ocular hypertension)
  Participants
    Open-angle glaucoma | 30 | 30 | 30 | 30 | 30 | 30 | 30 | 210
    Ocular hypertension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 12 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 12 months post-administration as assessed by liquid chromatography tandem mass spectrometry (LC-MS/MS)
Time Frame: month 12
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 1 (12-month Exchange)
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
ng/mL | 5.57 (3.02)

2. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 3 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 3 months post-administration as assessed by LC-MS/MS
Time Frame: month 3
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 2 (3-month Exchange)
Number analyzed (Participants) | 27
Number analyzed (eyes) | 27
ng/mL | 4.98 (2.50)

3. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 6 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 6 months post-administration as assessed by LC-MS/MS
Time Frame: month 6
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 3 (6-month Exchange)
Number analyzed (Participants) | 25
Number analyzed (eyes) | 25
ng/mL | 3.74 (2.22)

4. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 24 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 24 months post-administration as assessed by LC-MS/MS
Time Frame: month 24
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 4 (24-month Exchange)
Number analyzed (Participants) | 25
Number analyzed (eyes) | 25
ng/mL | 3.35 (1.51)

5. Primary Outcome: Travoprost Free Acid Concentration(ng/mL) in Aqueous Humor 21 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 21 months post-administration as assessed by LC-MS/MS
Time Frame: month 21
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 5 (21-month Exchange)
Number analyzed (Participants) | 27
Number analyzed (eyes) | 27
ng/mL | 3.80 (1.58)

6. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 18 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 18 months post-administration as assessed by LC-MS/MS
Time Frame: month 18
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Cohort 6 (18-month Exchange)
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
ng/mL | 2.22 (1.24)

7. Primary Outcome: Travoprost Free Acid Concentration (ng/mL) in Aqueous Humor 15 Months Post-administration
Description: concentration of travoprost free acid (ng/mL) in the aqueous humor 15 months post-administration as assessed by LC-MS/MS
Time Frame: month 15
Population: study eyes
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Groups:
- Cohort 7 15-month Exchange): Travoprost Intracameral Implant Exchanged at Month 15
  Travoprost Intracameral Implant exchanged at Month 15: intracameral implant containing travoprost 75 mcg implanted on Day 1 and exchanged at Month 15
Arm/Group | Cohort 7 15-month Exchange)
Number analyzed (Participants) | 28
Number analyzed (eyes) | 28
ng/mL | 2.03 (0.736)

8. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 12 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 12 months post-administration as assessed by high performance liquid chromatography (HPLC)
Time Frame: month 12
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: eyes
Arm/Group | Cohort 1 (12-month Exchange)
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
percentage of initial | 50.2 (6.58)

9. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 3 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 3 months post-administration as assessed by HPLC
Time Frame: month 3
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Error); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 2 (3-month Exchange)
Number analyzed (Participants) | 29
Number analyzed (explanted implants) | 29
percentage of initial | 78.8 (3.15)

10. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 6 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 6 months post-administration as assessed by HPLC
Time Frame: month 6
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 3 (6-month Exchange)
Number analyzed (Participants) | 28
Number analyzed (explanted implants) | 28
percentage of initial | 69.8 (8.51)

11. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 24 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 24 months post-administration as assessed by HPLC
Time Frame: month 24
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 4 (24-month Exchange)
Number analyzed (Participants) | 25
Number analyzed (explanted implants) | 25
percentage of initial | 16.3 (7.88)

12. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 21 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 21 months post-administration as assessed by HPLC
Time Frame: month 21
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 5 (21-month Exchange)
Number analyzed (Participants) | 27
Number analyzed (explanted implants) | 27
percentage of initial | 28.0 (5.76)

13. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 18 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 18 months post-administration as assessed by HPLC
Time Frame: month 18
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 6 (18-month Exchange)
Number analyzed (Participants) | 29
Number analyzed (explanted implants) | 29
percentage of initial | 34.8 (7.09)

14. Secondary Outcome: Percent Residual Travoprost in Explanted Implant 15 Months Post-administration
Description: percent of travoprost compared to baseline in explanted implant 15 months post-administration as assessed by HPLC
Time Frame: month 15
Population: explanted travoprost intracameral implants
Measure: Mean (Standard Deviation); unit: percentage of initial
Units Other Than Participants: explanted implants
Arm/Group | Cohort 7 (15-month Exchange)
Number analyzed (Participants) | 28
Number analyzed (explanted implants) | 28
percentage of initial | 38.6 (8.23)

ADVERSE EVENTS:
Time Frame: initial travoprost intracameral implant period plus 4 weeks post-exchange
Arm/Group | Cohort 1 (12-month Exchange) | Cohort 2 (3-month Exchange) | Cohort 3 (6-month Exchange) | Cohort 4 (24-month Exchange) | Cohort 5 (21-month Exchange) | Cohort 6 (18-month Exchange) | Cohort 7 (15-month Exchange)
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30 | 0/30 | 0/30 | 1/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/30 | 0/30 | 1/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 0/30 | 5/30 | 3/30 | 0/30 | 1/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (12-month Exchange) (N=30) | Cohort 2 (3-month Exchange) (N=30) | Cohort 3 (6-month Exchange) (N=30) | Cohort 4 (24-month Exchange) (N=30) | Cohort 5 (21-month Exchange) (N=30) | Cohort 6 (18-month Exchange) (N=30) | Cohort 7 (15-month Exchange) (N=30)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (12-month Exchange) (N=30) | Cohort 2 (3-month Exchange) (N=30) | Cohort 3 (6-month Exchange) (N=30) | Cohort 4 (24-month Exchange) (N=30) | Cohort 5 (21-month Exchange) (N=30) | Cohort 6 (18-month Exchange) (N=30) | Cohort 7 (15-month Exchange) (N=30)
Corona virus infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridodialysis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was open-label, non-randomized and conducted at a single site; however, the endpoints were objective and analyses of aqueous humor concentrations of travoprost free acid and of residual travoprost in explants were performed by a third party

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT06582732/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT06582732/SAP_001.pdf